CLINICAL TRIAL: NCT00624663
Title: A Double-Blind, Placebo-controlled Crossover Study to Assess the Pharmacokinetic Profile and the Physiological and Behavioral Effects of Repeat Rivastigmine (Exelon®) Administration in Young Healthy Male Volunteers
Brief Title: A Double-Blind, Placebo-controlled Crossover Study of Repeat Rivastigmine Administration in Healthy Male Volunteers
Acronym: RIVA-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Medical Corps, Israel Defense Force (Other)
Responsible Party: Jacob Atsmon, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TASMC-07-JA-234-CTIL; TRC 032/10058
Record Dates: First submitted 2007-10-30; First posted 2008-02-27 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2008-02

CONDITIONS: Rivastigmine Toxicity
Keywords: Rivastigmine, Repeated administration, Healthy Volunteers, organophosphate poisoning, protection, pharmacokinetics, behavioral effects
MeSH Terms: conditions — Organophosphate Poisoning | interventions — Rivastigmine; lactitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): (1 x 1.5 mg Exelon® Capsule (Novartis) + 1 x Placebo Capsule) X 2 per day, total of 5 intakes
  Interventions: Drug: Rivastigmine
- 2 (Active Comparator): (2 x 1.5 mg Exelon® Capsules) X 2 per day, total of 5 intakes
  Interventions: Drug: Rivastigmine
- 3 (Placebo Comparator): (2 x Placebo Capsules) X 2 per days, total of 5 intakes
  Interventions: Drug: Rivastigmine

INTERVENTIONS:
Drug: Rivastigmine — Administration 1 (A): 1 x 1.5 mg Exelon® Capsule (Novartis) + 1 x Placebo Capsule Administration 2 (B): 2 x 1.5 mg Exelon® Capsules (Novartis) Administration 3 (C): 2 x Placebo Capsules
  Other Names: Exelon® Capsules (Novartis)

SUMMARY:
Rivastigmine is a carbamate, approved by the FDA for the treatment of mild to moderate dementia associated with Alzheimer's and Parkinson's diseases. Studies conducted in the Israel Institute of Biological Research (IIBR) have yielded encouraging results in utilizing rivastigmine pre-treatment as an alternative to pyridostigmine in partially protecting against organophosphate poisoning, particularly protecting the central nervous system.

The target population for this indication may consist of otherwise healthy people (e.g. soldiers). Although the treatment regimen has not been established yet it is assumed, based on animal experiments, that rivastigmine is likely to be administered in repeated doses. In this setting, further evaluation of the drug's effects and pharmacokinetics in young healthy subjects is warranted.

The objectives of this study are: 1) To assess the safety and tolerability of repeated rivastigmine administration (1.5 mg and 3 mg) in young healthy male volunteers; 2) To determine the pharmacokinetic profile of rivastigmine (1.5 mg and 3 mg) following a single and multiple dose administrations; 3) To assess the extent of blood ChE inhibition following a single and multiple administrations of rivastigmine and 4) To correlate physiological and behavioral effects with blood rivastigmine concentrations and blood ChE inhibition in these subjects.

This double-blind, placebo-controlled study will be divided in 3 identical periods, preceded with a two-day initial training in performing cognitive performance tests. Each period will consist of in-house confinement for 5 days in which rivastigmine will be administered 5 times at an interval of 12 hours. During each period, each subject will receive either rivastigmine 1.5 mg X 5, or either rivastigmine 3.0 mg X 5 or placebo X 5. The treatment in each period will be randomly assigned in a crossover manner. Rivastigmine pharmacokinetics will and acetylcholinesterase inhibition will be assessed after the first and the last dose of each period and will be correlated with physiological and cognitive parameters: performance tests, visual functions, peak airway flow, saliva production (sialometry) and vital signs.

The emergence of adverse events will be monitored throughout the study

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian males between 18 and 40 years (inclusive) of age.
* No known history of significant neurological, renal, cardiovascular, respiratory (asthma), endocrinological, gastrointestinal, hematopoietic disease, neoplasm or any other clinically significant medical disorder, which in the investigator's judgment contraindicate administration of the study medications.
* Subjects within BMI 18-29 (inclusive) calculated as Weight (Kg)/Height (m)2.
* Non-smoking (by declaration) for a period of at least 6 months.
* No history of drug or alcohol abuse.
* Subjects with negative urinary drugs of abuse screen (Appendix 2) determined within 21 days of the start of the study.
* Negative HIV, Hepatitis B or Hepatitis C serology tests within 21 days of the first study session.
* Subjects must be able to adhere to the visit schedule and protocol requirements and be available to complete the study.
* Subjects must be fluent in Hebrew
* Subjects must satisfy a medical examiner about their fitness to participate in the study.
* Subjects must provide written informed consent to participate in the study.

Exclusion Criteria:

* • Known hypersensitivity to the drug, components or other carbamates.

  * History of or currently active asthma or chronic obstructive pulmonary disease.
  * History of or currently active cardiac arrhythmias such as bradycardia and sick sinus syndrome
  * History of urinary tract obstruction.
  * History of or currently active GI diseases such as peptic ulcer, GERD, bleeding or history of any GI surgery other than appendectomy or herniotomy, or with any gastrointestinal disorder likely to influence drug absorption, or with any history of anorexia, frequent nausea or emesis, regardless of etiology.
  * Significant abnormalities in screening physical exam
  * Significant abnormalities in clinical laboratory parameters (hematology, biochemistry, serology, urinalysis). Parameters to be measured are those shown in Appendix 2.
  * Significant abnormalities in ECG within 21 days of the start of the study.
  * Subjects with significant allergic response to other drugs.
  * Adherence (for whatever reason) to an abnormal diet during the 4 weeks prior to the study, or subjects with recent significant change in body weight.
  * Subjects who have taken anticholinergic or other drugs known to affect gastrointestinal motility within 7 days prior to the first dosing.
  * Use of any prescription or over-the-counter (OTC) medications, including vitamins and herbal or dietary supplements within 7 days prior to the first study dosing or during the study. Paracetamol for symptomatic relief of pain is allowed until 24 hours prior to the trial (see section 10.1).
  * Subjects who donated blood in the three months preceding the first study dosing or intend to make blood donation during the study, or within the three months following the study completion.
  * Subjects who received blood or plasma derivatives in the 3 months preceding the first study dosing.
  * Participation in another clinical trial with drugs within 3 months prior first study dosing.
  * Subjects with an inability to communicate well with the investigators and CRC staff (i.e., language problem, poor mental development or impaired cerebral performance).
  * Subjects that have difficulty fasting or consuming the standard meals that will be provided.
  * Subjects with any acute medical situation (e.g. acute infection) within 48 hours of study start, which is considered of significance by the Principal Investigator.
  * Subjects who are non-cooperative or unwilling to sign a consent form.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Physiological effects,Objective and subjective symptoms, Cognitive Performance tests | 5 weeks

SECONDARY OUTCOMES:
4. Pharmacokinetic parameters (Cmax, Tmax, AUCT, AUCI ) determined from plasma rivastigmine concentrations,Blood cholinesterase inhibition | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: JACOB ATSMON, MD, Principal Investigator — TASMC CLINICAL RESEARCH CENTER
Locations (2):
- Israel (2):
  - Tasmc Clinical Research Center, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv